CLINICAL TRIAL: NCT07098000
Title: The Role of Confocal Microscopy in Estimating Dupilumab Treatment Response for Moderate/Severe Atopic Dermatitis
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, LUIS DANIEL MAZZUOCCOLO, Head of Department of Dermatology, Hospital Italiano de Buenos Aires
Other Study IDs: 6955
Record Dates: First submitted 2025-07-03; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; reflectance confocal microscopy; dupilumab
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Dupilumab treated patients: Dupilumab treated patients
- Control: 10 healthy controls, five males and five females

SUMMARY:
Atopic dermatitis (AD) is recognized as the most prevalent chronic inflammatory skin disease across all age groups. The introduction of reflectance confocal microscopy (RCM) signifies a substantial leap forward in the non-invasive skin assessment at a cellular level. This advancement holds the potential to diminish the need for skin biopsies in diagnosing and monitoring skin diseases. Given the variability in the efficacy of systemic treatments for AD among patients, RCM emerges as an attractive tool for real-time monitoring of treatment response. This capability enables the treating physician to customize treatment approaches accordingly. There exists a lack of data concerning the subsurface characteristics of the skin explored with RCM before, during, and after dupilumab treatment in patients with moderate to severe AD.

Hypothesis: The characteristics of AD skin at the cellular level evaluated by RCM correlate with treatment response with dupilumab Overall objectives: To evaluate the association between skin characteristics assessed by basal RCM and changes in EASI and vIGA-AD scores at 24 weeks in individuals with mod/sev AD treated with dupilumab.

Methods: Prospective cohort study. Forty patients with mod/sev AD starting dupilumab will be enrolled. Basal and periodic clinimetry, PROs, and evaluation of the affected skin through RCM will be done.

Expected results: To describe RCM phenotypes of responders and not responders to dupilumab Impact: Offering the medical community a non-invasive tool to improve phenotypic characterization for tailoring clinical decisions. The investigators strongly believe this could mark the initial stride towards adopting personalized medicine, ultimately resulting in enhanced therapeutic selection, dosage precision, optimized intervals, increased patient adherence, and reducing need for skin biopsies, particularly in infants.

DETAILED DESCRIPTION:
Study Design and Setting

This is a prospective cohort study conducted at Hospital Italiano de Buenos Aires, a high-complexity, non-profit institution with a longstanding commitment to patient care, medical education, and research. The Department of Dermatology spans over 17 clinical sites and is one of the largest in Argentina, with 155,000 annual consultations and a strong focus on immune-mediated skin disorders, including atopic dermatitis (AD). The Division of Immune Skin Diseases includes 12 board-certified dermatologists specialized in managing complex inflammatory skin conditions. Our department actively participates in the Atopic Dermatitis Quality of Care Initiative and collaborates with local and international networks such as the Argentine Society of Dermatology, Pediatric Dermatology Society, and Project ECHO® AD group.

Study Population and Recruitment Strategy

The study will enroll patients from the Buenos Aires Metropolitan Area (population ~14 million), where an estimated 3% of adults and 5% of children are affected by AD, with moderate-to-severe cases representing approximately 0.3%-0.5%. Dermatologists and allergists across all sectors-public, private, and social security-will be invited to refer eligible patients prior to dupilumab treatment initiation. Inclusion will not be restricted by insurance status or care setting, ensuring demographic and socioeconomic diversity.

Study Procedures

Patients will be referred to Hospital Italiano, where the study team will conduct consent and baseline evaluations. Study duration is up to 48 weeks, including four visits: baseline, week 12 and week 24. Systemic treatment will be prescribed independently by the referring physician, allowing the study to observe real-world therapeutic strategies. The coordinating center will manage clinimetric assessments, patient-reported outcomes (PROs), and imaging.

Baseline Assessments:

Demographics and medical history. Clinimetry: vIGA-AD, EASI, BSA, SCORAD, PGIS, PGIC. PROs: PP-NRS, SP-NRS, Sleep-NRS, POEM, ADCT, DLQI. Documentation of prescribed treatment: molecule, route, dose, schedule. RCM imaging of selected lesions (trunk, limbs, face), excluding hyperkeratotic or eroded acral lesions.

RCM Imaging Protocol:

Equipment: Vivascope 1500 and 3000 (Caliber ID). Mosaic acquisition (5x5 mm) at four skin depths: stratum corneum, stratum spinosum, dermoepidermal junction, and superficial dermis.

Stacked images collected from the corneal layer to ~250 μm depth. Facial lesions will be imaged with the handheld Vivascope 3000 when needed. Images stored in a secured, structured database.

Follow-Up Visits (Weeks 12 and 24):

Repeat clinimetry and PRO assessments. Treatment adherence and adverse event monitoring. Repeat RCM imaging on the same anatomical sites.

Predictive and Descriptive Variables:

RCM features: parakeratosis, hyperkeratosis, spongiosis, vesicles, acanthosis, exocytosis, non-edged dermal papillae, DEJ morphology, vascular dilation, dermal infiltration, melanophages.

Clinical: phenotype (e.g., classical, nummular, generalized lichenoid), comorbidities, prior therapies, IgE levels, family history.

Sample Size and Sampling Strategy

This exploratory study does not have a formal sample size estimation. The investigators expect to include 40 consecutive patients on dupilumab therapy, at least ten patients with the main phenotypes:

1. Classical: Lichenified/exudative flexural dermatitis, almost always associated with head-and-neck eczema and hand eczema
2. Generalized eczema with a lichenoid pattern: lichenification, excoriations, crusts, and xerosis
3. Nummular eczema with round, inflamed sores.

Statistical Analysis

Descriptive statistics will include frequencies for categorical variables and medians with interquartile ranges for continuous variables.

Primary analysis: Linear regression using the change (Δ) in EASI and vIGA-AD from baseline to week 24 as outcomes; baseline RCM features as predictors.

Secondary analysis: Logistic regression for binary clinical responses (e.g., achieving EASI-75), reporting odds ratios (ORs) with 95% confidence intervals (CIs).

All analyses will be conducted using STATA v14.1.

ELIGIBILITY:
Inclusion Criteria:

* ≥6 months of age.
* Diagnosis of AD based on Hanifin and Rajka criteria.
* Moderate-to-severe AD defined by: EASI >16, BSA >10%, SCORAD >25, or vIGA-AD 3-4.
* Starting dupilumab for AD indicated and initiated by the attending physician.
* Signed informed consent or assent with guardian approval.
* In those with previous systemic treatment (jaki, oral steroids, methotrexate and phototherapy), a predefined wash-out time of 4 weeks must be guaranteed.

Exclusion Criteria:

* Inability to comply with study procedures.
* Refusal to provide informed consent.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will enroll patients from the Buenos Aires Metropolitan Area (population ~14 million), where an estimated 3% of adults and 5% of children are affected by AD, with moderate-to-severe cases representing approximately 0.3%-0.5%. Dermatologists and allergists across all sectors-public, private, and social security-will be invited to refer eligible patients prior to dupilumab treatment initiation. Inclusion will not be restricted by insurance status or care setting, ensuring demographic and socioeconomic diversity.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2025-12-12 (Estimated); Study Completion 2026-04-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between baseline RCM features and change in EASI score at week 24 | Baseline and week 24
  The correlation between baseline reflectance confocal microscopy (RCM) features (e.g., spongiosis, inflammatory cell infiltrate, disarrayed epidermis, changes in the dermoepidermal junction) and the change in Eczema Area and Severity Index (EASI) from baseline to week 24 will be assessed.
  Measurement Tool: Eczema Area and Severity Index (EASI) Unit of Measure: Change in EASI score (continuous variable)
Correlation between baseline RCM features and change in vIGA-AD score at week 24 | Baseline and week 24
  The correlation between baseline RCM features and the change in validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) from baseline to week 24 will be assessed.
  Measurement Tool: Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) Unit of Measure: Change in vIGA-AD score (ordinal scale 0-4)

SECONDARY OUTCOMES:
Predictive value of baseline RCM features for achieving EASI-75 at week 24 | From enrollment to week 24
  The association between baseline reflectance confocal microscopy (RCM) features (e.g., spongiosis, inflammatory infiltrate, disarrayed epidermis, changes in the dermoepidermal junction) and achieving at least 75% improvement in Eczema Area and Severity Index (EASI-75) at week 24 will be evaluated.
  Measurement Tool: Eczema Area and Severity Index (EASI) Unit of Measure: % of participants achieving EASI-75
Predictive value of baseline RCM features for achieving vIGA-AD 0 or 1 at week 24 | From enrollment to week 24
  The association between baseline RCM features and achieving a score of 0 (clear) or 1 (almost clear) in the validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) at week 24 will be evaluated.
  Measurement Tool: Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) Unit of Measure: % of participants achieving vIGA-AD 0 or 1
Predictive value of baseline RCM features for achieving EASI <10 at week 24 | From enrollment to week 24
  The association between baseline RCM features and achieving an EASI score <10 at week 24 will be evaluated.
  Measurement Tool: Eczema Area and Severity Index (EASI) Unit of Measure: % of participants with EASI <10
Correlation between baseline RCM features and change in SCORAD at week 24 | From enrollment to week 24
  The correlation between baseline reflectance confocal microscopy (RCM) features and change in SCORAD (Scoring Atopic Dermatitis) from baseline to week 24 will be assessed.
  Measurement Tool: SCORAD index Unit of Measure: Change in SCORAD score (continuous variable)
Correlation between baseline RCM features and change in BSA affected at week 24 | From enrollment to week 24
  The correlation between baseline RCM features and change in Body Surface Area (BSA) affected by atopic dermatitis from baseline to week 24 will be assessed.
  Measurement Tool: Clinician-estimated BSA Unit of Measure: Change in % BSA affected
Correlation between baseline RCM features and change in Patient Global Impression of Severity (PGIS) at week 24 | From enrollment to week 24
  The correlation between baseline RCM features and change in PGIS scores from baseline to week 24 will be assessed.
  Measurement Tool: Patient Global Impression of Severity (PGIS) Unit of Measure: Change in PGIS score (ordinal scale)
Correlation between baseline RCM features and Patient Global Impression of Change (PGIC) at week 24 | Week 24
  The correlation between baseline RCM features and PGIC score at week 24 will be assessed.
  Measurement Tool: Patient Global Impression of Change (PGIC) Unit of Measure: PGIC score at week 24 (ordinal scale)
Correlation between baseline RCM features and change in peak pruritus NRS at week 24 | From enrollment to week 24
  The correlation between baseline RCM features and change in peak pruritus Numeric Rating Scale (NRS) score from baseline to week 24 will be assessed.
  Measurement Tool: Peak Pruritus NRS (0-10) Unit of Measure: Change in NRS score (continuous variable)
Correlation between baseline RCM features and change in POEM score at week 24 | From enrollment to week 24
  The correlation between baseline RCM features and change in Patient-Oriented Eczema Measure (POEM) from baseline to week 24 will be assessed.
  Measurement Tool: POEM questionnaire Unit of Measure: Change in POEM score (continuous variable)
Correlation between baseline RCM features and change in Atopic Dermatitis Control Tool (ADCT) score at week 24 | From enrollment to week 24
  The correlation between baseline RCM features and change in ADCT score from baseline to week 24 will be assessed.
  Measurement Tool: Atopic Dermatitis Control Tool (ADCT) Unit of Measure: Change in ADCT score (continuous variable)
Correlation between baseline RCM features and change in Dermatology Life Quality Index (DLQI) at week 24 | From enrollment to week 24
  The correlation between baseline RCM features and change in DLQI score from baseline to week 24 will be assessed.
  Measurement Tool: Dermatology Life Quality Index (DLQI) Unit of Measure: Change in DLQI score (continuous variable)
Association between clinical phenotype and achievement of EASI-75 at week 24 | From enrollment to week 24
  The association between baseline clinical phenotype and achieving at least 75% improvement in EASI score (EASI-75) at week 24 will be assessed.
  Measurement Tool: Eczema Area and Severity Index (EASI) Unit of Measure: % of participants achieving EASI-75
Association between age of onset and achievement of EASI-75 at week 24 | From enrollment to week 24
  The association between age at onset of atopic dermatitis and achieving EASI-75 at week 24 will be evaluated.
  Measurement Tool: EASI Unit of Measure: % of participants achieving EASI-75
Association between family history of atopic disease and achievement of EASI-75 at week 24 | From enrollment to week 24
  The association between family history of atopic disease and the likelihood of achieving EASI-75 at week 24 will be assessed.
  Measurement Tool: EASI Unit of Measure: % of participants achieving EASI-75
Association between previous treatment failures and achievement of EASI-75 at week 24 | From enrollment to week 24
  The association between prior failure of topical or systemic treatments and achieving EASI-75 at week 24 will be evaluated.
  Measurement Tool: EASI Unit of Measure: % of participants achieving EASI-75
Incidence and severity of adverse events during treatment | From enrollment to week 24
  Adverse events occurring during the 24-week treatment period will be recorded and classified by severity according to the Common Terminology Criteria for Adverse Events (CTCAE).
  Measurement Tool: CTCAE v5.0 Unit of Measure: Number of adverse events per CTCAE grade
Rate of patient adherence to treatment | From enrollment to week 24
  Patient adherence will be evaluated as the percentage of prescribed doses (topical and/or systemic) that were effectively administered over the 24-week period.
  Measurement Tool: Patient and/or caregiver diary Unit of Measure: % of prescribed doses taken
Frequency of treatment modifications (interruptions or switching) | From enrollment to week 24
  The number and proportion of patients requiring treatment interruption, discontinuation, or change of therapy will be recorded to assess feasibility of the intervention.
  Measurement Tool: Study medication records Unit of Measure: % of participants with treatment modifications
Change in composite RCM score from baseline to week 24 | Baseline and week 24
  A composite RCM score (based on presence of spongiosis, inflammatory infiltrate, epidermal disarray, and DEJ abnormalities) will be calculated at baseline and week 24. Mean changes in score will be analyzed across the cohort and by clinical response (EASI-75).
  Measurement Tool: Investigator-assessed composite RCM score (0-12) Unit of Measure: Mean change in score (continuous variable)
Difference in composite RCM score between AD patients and healthy controls | Time Frame: Baseline only
  A composite reflectance confocal microscopy (RCM) score will be calculated at baseline for each participant based on the presence and severity of four predefined imaging features: spongiosis, inflammatory cell infiltrate, epidermal disarray, and dermoepidermal junction (DEJ) abnormalities. Mean scores will be compared between patients with atopic dermatitis and age-matched healthy controls to identify structural markers of disease.
  Measurement Tool: Investigator-assessed composite RCM score (0-12) Unit of Measure: Mean composite score (continuous variable)

CONTACTS AND LOCATIONS:
Overall Officials: Luis D Mazzuoccolo, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yew YW, Dinish US, Choi ECE, Bi R, Ho CJH, Dev K, Li X, Attia ABE, Wong MKW, Balasundaram G, Ntziachristos V, Olivo M, Thng STG. Investigation of morphological, vascular and biochemical changes in the skin of an atopic dermatitis (AD) patient in response to dupilumab using raster scanning optoacoustic mesoscopy (RSOM) and handheld confocal Raman spectroscopy (CRS). J Dermatol Sci. 2019 Sep;95(3):123-125. doi: 10.1016/j.jdermsci.2019.07.003. Epub 2019 Jul 12. No abstract available. PMID 31558224
- [Background] Csuka EA, Ward SC, Ekelem C, Csuka DA, Ardigo M, Mesinkovska NA. Reflectance Confocal Microscopy, Optical Coherence Tomography, and Multiphoton Microscopy in Inflammatory Skin Disease Diagnosis. Lasers Surg Med. 2021 Aug;53(6):776-797. doi: 10.1002/lsm.23386. Epub 2021 Feb 1. PMID 33527483
- [Background] Berdyshev E, Goleva E, Bissonnette R, Bronova I, Bronoff AS, Richers BN, Garcia S, Ramirez-Gama M, Taylor P, Praestgaard A, Agueusop I, Jurvilliers P, Boguniewicz M, Levit NA, Rossi AB, Zhang A, Leung DYM. Dupilumab significantly improves skin barrier function in patients with moderate-to-severe atopic dermatitis. Allergy. 2022 Nov;77(11):3388-3397. doi: 10.1111/all.15432. Epub 2022 Jul 21. PMID 35815904
- [Background] Beck LA, Deleuran M, Bissonnette R, de Bruin-Weller M, Galus R, Nakahara T, Seo SJ, Khokhar FA, Vakil J, Xiao J, Marco AR, Levit NA, O'Malley JT, Shabbir A. Dupilumab Provides Acceptable Safety and Sustained Efficacy for up to 4 Years in an Open-Label Study of Adults with Moderate-to-Severe Atopic Dermatitis. Am J Clin Dermatol. 2022 May;23(3):393-408. doi: 10.1007/s40257-022-00685-0. Epub 2022 May 3. PMID 35503163
- [Background] Beck LA, Cork MJ, Amagai M, De Benedetto A, Kabashima K, Hamilton JD, Rossi AB. Type 2 Inflammation Contributes to Skin Barrier Dysfunction in Atopic Dermatitis. JID Innov. 2022 Apr 26;2(5):100131. doi: 10.1016/j.xjidi.2022.100131. eCollection 2022 Sep. PMID 36059592
- [Background] Antonietti C, Angles MV, Giachetti A, Diaz MS, Gloser D, Juszkiewicz E, Parrales Villacreses M, Mazzuoccolo L, Parisi C. Atopic dermatitis in children and adolescents seen at a general hospital in the City of Buenos Aires. Arch Argent Pediatr. 2023 Jun 1;121(3):e202202639. doi: 10.5546/aap.2022-02639.eng. Epub 2022 Dec 1. English, Spanish. PMID 36445075
- [Background] Angles MV, Antonietti CA, Torre AC, Juszkiewicz Franze E, Mazzuoccolo LD, Parisi CAS. Prevalence of atopic dermatitis in adults. An Bras Dermatol. 2022 Jan-Feb;97(1):107-109. doi: 10.1016/j.abd.2020.10.016. Epub 2021 Nov 26. No abstract available. PMID 34839985

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-09): https://cdn.clinicaltrials.gov/large-docs/00/NCT07098000/Prot_SAP_000.pdf